CLINICAL TRIAL: NCT05032378
Title: Efficacy of a Motion Sensor and Feedback System to Refine Movements of People With Acquired Neurological Injury: A Series of Case Studies
Brief Title: Motion Sensor and Feedback System Efficacy to Refine Movements After Injury
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: PantherTec (Industry)
Collaborators: Quality Living, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: KAT
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injuries; Stroke; Acquired Brain Injury; Movement Disorders
Keywords: efficacy; Treatment
MeSH Terms: conditions — Spinal Cord Injuries; Stroke; Brain Injuries; Movement Disorders | interventions — Occupational Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with movement disorders: Adults with acquired movement disorders secondary to neurological injury.
  Interventions: Behavioral: Kinesthetic Awareness Training
- Professionals: Professionals providing physical or occupational therapy to participants with acquired movements disorders.
  Interventions: Behavioral: Provision of KAT-assisted physical or occupational therapy

INTERVENTIONS:
Behavioral: Kinesthetic Awareness Training — One physical or occupational therapy session per week for 8 weeks during which the participant with disordered movement will attempt to perform desired movements while wearing the KAT device
  Other Names: KAT
  Groups: People with movement disorders
Behavioral: Provision of KAT-assisted physical or occupational therapy — Physical or occupational therapy professionals will provide one KAT-assisted therapy session per week for 8 weeks to one or more participants with movement disorder.
  Groups: Professionals

SUMMARY:
The purpose of these case studies is to determine the efficacy of the Kinesthetic Awareness Training (KAT) device in facilitating the restoration of desired movement patterns when people with acquired central nervous system damage perform functional activities such as walking, transitioning from one position to another, or reaching with the arms.

DETAILED DESCRIPTION:
People with acquired neurological disorders often exhibit impaired movement patterns when performing functional activities such as walking, standing up from a seated position, and reaching for objects. Re-establishing normal movement patterns is an essential part of rehabilitation; however, achievement of this typically requires thousands of accurate movement repetitions. Only through this repetition can a person benefit from the inherent neuroplasticity of the nervous system to make restored patterns habitual.

Sensory and/or proprioceptive problems may limit a person's awareness of ways in which abnormal movement patterns differ from desired ones. Because of these problems, provision of external feedback in the form of verbal comments, physical repositioning of the limbs by another person, or other auditory or haptic cues is critical. As a general rule, a person benefits most when provided with precise feedback about the position of body parts when he/she is actively engaged in performing a desired movement. As such, the linking of motion sensors programmed to detect achievement of a target position with immediate auditory (i.e., beeps) and/or haptic (i.e., vibrations) feedback has the potential to be a powerful treatment tool.

The Kinesthetic Awareness Training (KAT) device developed by PantherTec is a wearable, motion capture system that can be programmed to detect and provide immediate auditory and/or haptic feedback when a person moves a specified body part to a target position during performance of a functional sequence of movements. Each time a person replicates the desired movement, the device either begins emitting or ceases emitting beeps and/or vibrations-as specified during programming-to indicate achievement of the correct position. Adjustment of the sensitivity (i.e., margin of error per target value) allows for specification of how close a performed movement must be to the target position to elicit feedback.

PantherTec has made a prototype of the KAT device available to Quality Living, Inc. (QLI) for feasibility testing and exploration of possible applications with people with movement impairments resulting from acquired neurological injury. The purpose of the proposed case studies is to determine the efficacy of the KAT device in facilitating the restoration of desired movement patterns when people with acquired central nervous system damage perform functional activities such as walking, transitioning from one position to another, or reaching with the arms.

ELIGIBILITY:
Inclusion Criteria:

* For participants with movement disorders:

  * Between 16 and 70 years of age
  * Has an acquired movement disorder secondary to neurological injury
  * Understands English sufficiently to follow simple commands
  * Is a current resident of Quality Living, Inc.
* For professionals:

  * Over 19 years of age
  * A physical therapy or occupational therapy staff member employed by Quality Living, Inc.
  * Has used the KAT device to provide treatment to a participant with a movement disorder

Exclusion Criteria:

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Current residents of Quality Living, Inc., who are receiving treatment for an acquired movement disorder.
  Current staff of Quality Living, Inc., who are providing physical or occupational therapy treatment to a participant with an acquired movement disorder.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scaling (GAS) in rehabilitation | completion of 8-week treatment period
  The GAS uses a 5-point rating scale to describe the extent of a participant's goal achievement. Scores for each attainment goal range from -2 (much worse than expected) to +2 (much better than expected). The composite GAS (the sum of attainment levels x the relative weight for each goal) is transformed into a standardized measure or T score with a mean of 50 and standard deviation of 10.
System Usability Scale (SUS) | completion of 8-week treatment provision period
  The SUS is a feasibility rating scale for that will be used by professional participants to evaluate the KAT device. It includes 10 items with 5 response options ranging from 1 (strongly disagree) to 5 (strongly agree). Scores for odd-numbered items on the scale are calculated by subtracting 1 from the user's rating; scores for even-numbered items on the scale are calculated by subtracting the user's response from 5. This scales all values from 0 to 4, with four being the most positive response. Summing the converted scores and multiplying by 2.5 yields a score between 0 and 100, with 100 being the most positive score.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hux, Ph.D., Principal Investigator — Quality Living, Inc.
Locations (1):
- Quality Living, Inc., Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No